CLINICAL TRIAL: NCT04796961
Title: Promoting Evidenced-Based Tobacco Smoking Cessation Treatment in Community Mental Health Clinics
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00231836; 1P50MH115842-01 (NIH)
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation Intervention (Other): All participants will receive the implementation intervention.
  Interventions: Other: Implementation Intervention

INTERVENTIONS:
Other: Implementation Intervention — The implementation intervention involves training, coaching, expert consultation, organizational strategy meetings.

SUMMARY:
This pilot study will examine whether an implementation intervention will improve delivery of evidence-based treatment for tobacco smoking cessation for patients in community mental health clinics.

DETAILED DESCRIPTION:
In this pilot study, the investigators will work with community mental health clinical and pilot test an implementation intervention to improve mental health providers' delivery of evidence-based tobacco smoking cessation treatment in community mental health clinics.

ELIGIBILITY:
Inclusion Criteria:

* study population: community mental health clinic staff and providers

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Daumit, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dickerson F, Goldsholl S, Yuan CT, Dalcin A, Eidman B, Minahan E, Gennusa Rd JV, Mace E, Cullen B, Evins AE, Cather C, Wang NY, McGinty EM, Daumit GL. Promoting Evidence-Based Tobacco Cessation Treatment in Community Mental Health Clinics: Protocol for a Prepost Intervention Study. JMIR Res Protoc. 2023 May 12;12:e44787. doi: 10.2196/44787. PMID 37171851

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mental health clinic staff (providers and prescribers) were recruited from 5 mental health clinics.
Pre-assignment Details: Ninety-one mental health clinic staff (providers and prescribers) were enrolled in the study. The mental health clinics had 6,011 clients with data that were included in the analysis.
Units Other Than Participants: Clinics
Period: Overall Study
Arm/Group | Implementation Intervention
Started | 91; 5 Clinics
Mental Health Clinic Clients (Not Enrolled) | 6011; 5 Clinics
Completed | 68; 5 Clinics
Not Completed | 23; 0 Clinics
Not completed — Lost to Follow-up | 10
Not completed — Withdrawal by Subject | 3
Not completed — Left Organization | 10

BASELINE CHARACTERISTICS:
Arm/Group | Implementation Intervention
Number analyzed (Participants) | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 81
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.0 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 80
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 65
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 91
Staff Role [Count of Participants; unit: Participants] — Role of the staff member as it relates to delivery of the evidence-based practice intervention.
  Participants
    Counseling Provider | 54
    Prescriber | 37

OUTCOME MEASURES:

1. Primary Outcome: Provider (Staff) Knowledge of Smoking Cessation Treatment as Assessed by a 16-item Scale
Description: Knowledge of evidence-based smoking cessation treatment: 16-item scale developed by our team. Items are true/false and score reflects number answered correctly. Average score range 0-16 with a higher score signifies an increased knowledge of smoking cessation treatment.
Time Frame: Baseline, 12 months
Population: Staff with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implementation Intervention
Number analyzed (Participants) | 90
score on a scale
  Baseline | 13.8 (1.4)
  12 months | 14.2 (1.2)
Statistical Analysis 1: Comparison: Implementation Intervention; Test type: Superiority; Mean Difference (Net) = 0.4, 95% CI 2-sided [0.1 to 0.7]

2. Primary Outcome: Provider Self-efficacy to Deliver Evidence-based Smoking Cessation Treatment
Description: Self-efficacy for a four components of the smoking cessation intervention were evaluated using an instrument adapted from Compeau and Higgins' task-focused self-efficacy scale. Responses for items are on a Likert scale of 1-10. Average score range 1-10 and higher scores signify greater self-efficacy for the smoking cessation task.
Time Frame: Baseline, 12 months
Population: Staff with data collected analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Counseling Providers: Consented and enrolled staff participants at mental health organizations delivered smoking cessation counseling.
- Prescribers: Consented and enrolled staff participants at mental health organizations who prescribe medications
Arm/Group | Counseling Providers | Prescribers
Number analyzed (Participants) | 53 | 37
score on a scale
  Smoking Screening - Baseline | 7.1 (2) | 6.6 (2.9)
  Smoking Screening - 12 Months | 7.2 (2.2) | 7.2 (2.6)
  Readiness to Quit Assessment - Baseline | 6.7 (2.1) | 6.1 (3.2)
  Readiness to Quit Assessment - 12 Months | 7.3 (2.1) | 6.6 (3.2)
  Smoking Cessation Counseling - Baseline: number analyzed (Participants) | 53 | 0
  Smoking Cessation Counseling - Baseline | 5.5 (2.8) |
  Smoking Cessation Counseling - 12 Months: number analyzed (Participants) | 53 | 0
  Smoking Cessation Counseling - 12 Months | 7.0 (2.1) |
  Smoking Cessation Pharmacotherapy - Baseline: number analyzed (Participants) | 0 | 37
  Smoking Cessation Pharmacotherapy - Baseline |  | 6.2 (2.8)
  Smoking Cessation Pharmacotherapy - 12 Months: number analyzed (Participants) | 0 | 37
  Smoking Cessation Pharmacotherapy - 12 Months |  | 7.0 (2.9)
Statistical Analysis 1: Comparison: Counseling Providers vs Prescribers; smoking screening; Test type: Superiority; Mean Difference (Net) = 0.5, 95% CI 2-sided [-0.1 to 1.1]
Statistical Analysis 2: Comparison: Counseling Providers vs Prescribers; readiness to quit assessments; Test type: Superiority; Mean Difference (Net) = 0.6, 95% CI 2-sided [-0.1 to 1.2]
Statistical Analysis 3: Comparison: Counseling Providers; smoking cessation counseling; Test type: Superiority; Mean Difference (Net) = 1.4, 95% CI 2-sided [0.8 to 2.0]
Statistical Analysis 4: Comparison: Prescribers; smoking cessation pharmacotherapy; Test type: Superiority; Mean Difference (Net) = 0.6, 95% CI 2-sided [-0.5 to 1.7]

3. Secondary Outcome: Number of Clients Recieved Smoking Status Assessment
Description: Assessment of smoking status measured by clinic documentation during client visits with the number below indicating the number of clients who had a smoking status assessment during the 12 month study period.
Time Frame: Baseline through 12 months
Population: Mental health clinic clients
Measure: Count of Participants; unit: Participants
Arm/Group | Implementation Intervention
Number analyzed (Participants) | 6011
Participants | 3406

4. Secondary Outcome: Number of Clients Willing to Quit Smoking That Received a Willingness to Quit Assessment
Description: Assessment of willingness to quit measured by clinic documentation during client visits, with the number below indicating the number of clients who reported smoking during a smoking status assessment who had a willingness to quit assessment during the 12 month study period.
Time Frame: Baseline through 12 months
Population: Clients who had a smoking status assessment collected where they reported smoking during the study period were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Implementation Intervention
Number analyzed (Participants) | 1469
Participants | 1192

5. Secondary Outcome: Number of Clients Interested in Quitting Smoking Who Received Smoking Cessation Behavioral Counseling
Description: Receipt of behavioral counseling measured by clinic documentation during client visits, with the number below indicating the number of clients interested in quitting smoking that reported smoking during a smoking status assessment who staff reported as receiving behavioral counseling during the 12 months study period.
  Data is reported in two groups based upon whether the client had a recorded interest in quitting smoking or not, and only includes clients who reported smoking at some point during the study period. Clients can be reported in both groups if they responded differently to this question at two points over the course of the 12 months.
Time Frame: Baseline through 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Implementation Intervention
Number analyzed (Participants) | 1469
Participants
  Client Smokers Reported Interest in Quitting: number analyzed (Participants) | 644
  Client Smokers Reported Interest in Quitting | 529
  Clients Not Reported Interest In Quitting Smoking: number analyzed (Participants) | 1085
  Clients Not Reported Interest In Quitting Smoking | 759

6. Secondary Outcome: Number of Clients Interested in Quitting Smoking That Received Smoking Cessation Pharmacotherapy
Description: Measured by clinic documentation during client visits with the number below indicating the number of clients interested in quitting smoking, that reported smoking during a smoking status assessment who staff reported as receiving smoking cessation pharmacotherapy during the 12 months study period.
  Clients can be reported in both groups (Interested in quitting, not interested in quitting) if they responded differently to this question at two points over the course of the 12 months.
Time Frame: Baseline through 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Implementation Intervention
Number analyzed (Participants) | 1469
Participants
  Client Smokers Reported Interest in Quitting: number analyzed (Participants) | 644
  Client Smokers Reported Interest in Quitting | 232
  Client Smokers Not Reported Interest in Quitting: number analyzed (Participants) | 1085
  Client Smokers Not Reported Interest in Quitting | 173

7. Secondary Outcome: Acceptability of Evidence-based Practices Based on Adaptation of Acceptability of Intervention Measure
Description: An adaptation of the Acceptability of Intervention Measure was used. Each of the items will be measured on a 5-point Likert scale, where 1=completely disagree and 5=completely agree. An average score is calculated by summing responses across all four items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies greater acceptability.
Time Frame: Post Training (up to 2 weeks), 12 months
Population: Staff with data collected, analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implementation Intervention
Number analyzed (Participants) | 66
score on a scale
  Post Training | 4.1 (0.5)
  12 Months | 4.0 (0.7)

8. Secondary Outcome: Appropriateness of Evidence-based Practices Based on Adaptation of the Intervention Appropriateness Measure
Description: An adaptation of the Intervention Appropriateness Measure was used. Each of the items will be measured on a 5-point Likert scale, where 1=completely disagree and 5=completely agree. An average score is calculated by summing responses across all four items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies greater appropriateness.
Time Frame: Post Training (up to 2 weeks), 12 Months
Population: Staff with data collected, analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implementation Intervention
Number analyzed (Participants) | 66
score on a scale
  Post Training | 4.2 (0.5)
  12 Months | 4.1 (0.7)

9. Secondary Outcome: Feasibility of Evidence-based Practices Based on Adaptation of the Feasibility of Intervention Measure
Description: An adaptation of the Feasibility of Intervention Measure was used. Each of the items will be measured on a 5-point Likert scale, where 1=completely disagree and 5=completely agree. An average score is calculated by summing responses across all four items and dividing by the total number of items. The average score ranges from 1-5. A higher score signifies greater feasibility.
Time Frame: Post Training (up to 2 weeks), 12 Months
Population: Staff with data collected, analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implementation Intervention
Number analyzed (Participants) | 66
score on a scale
  Post Training | 4.1 (0.5)
  12 Months | 4.0 (0.7)

10. Secondary Outcome: Acceptability of Implementation Intervention Based on Adaptation of Acceptability of Intervention Measure
Description: as for outcome 7
Time Frame: Post Training (up to 2 weeks), 12 Months
Population: Staff with data collected, analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implementation Intervention
Number analyzed (Participants) | 66
score on a scale
  Post Training | 4.1 (0.6)
  12 Months | 3.9 (0.7)

11. Secondary Outcome: Appropriateness of Implementation Intervention Based on Adaptation of the Intervention Appropriateness Measure
Description: as for outcome 8
Time Frame: Post Training (up to 2 weeks), 12 Months
Population: Staff with data collected, analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implementation Intervention
Number analyzed (Participants) | 66
score on a scale
  Post Training | 4.1 (0.6)
  12 Months | 3.9 (0.7)

12. Secondary Outcome: Feasibility of Implementation Intervention Based on Adaptation of the Feasibility of Intervention Measure
Description: as for outcome 9
Time Frame: Post Training (up to 2 weeks), 12 Months
Population: Staff with data collected, analyzed under modeling approach.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implementation Intervention
Number analyzed (Participants) | 66
score on a scale
  Post Training | 4.0 (0.7)
  12 Months | 3.9 (0.7)

13. Other Pre Specified Outcome: Change in Tobacco Smoking Abstinence
Description: 7-day patient abstinence reported in medical record
Time Frame: Baseline, 12 Months
Population: Information data source was the health record and this data was not present routinely. When available the data appeared not to be valid.
Arm/Group | Implementation Intervention
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse Events Not Collected
Arm/Group | Implementation Intervention
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/61/NCT04796961/Prot_SAP_000.pdf